CLINICAL TRIAL: NCT07191197
Title: New Semantic Learning in Patients With Selective Brain Lesions in Temporal Regions: a Behavioural and MRI Study
Brief Title: How do Patients With Amnesia Acquire New Knowledge?
Acronym: ASSAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/23/0377
Record Dates: First submitted 2025-08-25; First posted 2025-09-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Amnesia; Memory Disorder
Keywords: Learning; Semantic memory; Hippocampus; Temporal pole
MeSH Terms: conditions — Amnesia; Memory Disorders | interventions — Psychometrics

STUDY DESIGN:
Intervention Model Description: sectional, experimental, comparative, bicentric study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Learning abilities for Patients with an amnesic syndrome (Experimental): 1 MRI session, 2 cognitive research tasks of semantic learning, and neuropsychological assessment.
  Interventions: Other: MRI; Other: Psychometric
- Healthy controls (Active Comparator): To allow multiple pairing for each patient, a group of 120 healthy controls aged between 18 to 70 years old will be recruited. Thus, it will be possible to compare one given patient to a group of 40 aged-matched subjects.
  All healthy volunteers will undergo the same intervention as the patients :
  1 MRI session, 2 cognitive research tasks of semantic learning, neuropsychological assessment.
  Interventions: Other: MRI; Other: Psychometric

INTERVENTIONS:
Other: MRI — structural and functional resting state MRI
Other: Psychometric — 2 cognitive research tasks of semantic learning and neuropsychological assessment

SUMMARY:
THE STUDY AIMS to constitute the largest group of patients with major memory impairment resulting from various etiology and specific lesions of the medial temporal lobe (MTL) and use a combined psychometric and neuroimaging approach to study the factors allowing these patients to successfully learn new semantic information.

DETAILED DESCRIPTION:
The preservation of learning abilities is an essential aspect in the implementation of cognitive rehabilitation programs for patients with an amnesic syndrome. Particularly disabled on a daily basis, these patients have significant difficulties in coping with the demands of work and family life. Data from previous case studies attest to the ability of these patients to rely on preserved cognitive systems to learn new semantic information. However, the procedures for the acquisition of new information are sometimes long, not optimal and the clinical factors, that can influence it, are poorly identified. In addition, the brain networks necessary for such learning are still debated. In order to better understand the cognitive mechanisms and brain networks that underlie the ability to learn new semantic information, the research aims to study a group of patients with major memory impairment following medial temporal lobe lesions of various etiologies (non-degenerative). The study will use a combined psychometric and neuroimaging approach to identify the factors that enable these patients to successfully learn new semantic information.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years
* Living in France since less than 20 years, being able to understand the French language, and have basic cultural knowledge as evaluated in classical clinical consultation
* Written agreement to participate in the study
* Intellectual capacities compatible with the cognitive tasks and signing of consent
* Affiliation to the French social security system
* For patients: bilateral brain lesion of the medial temporal lobe or the extended hippocampal system

Exclusion Criteria:

* Subjects under the age of 18 or over 70
* Contraindications for MRI (examples: wearers of a pacemaker or cardiac defibrillator, implanted equipment activated by an electrical, magnetic or mechanical system, wearers of haemostatic clips for intracerebral aneurysms or carotid arteries, wearers of orthopedic implants, claustrophobic)
* Refusal to be informed of an anomaly detected during the MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Performance on Fast-Mapping semantic learning task | Baseline
  * MRI measures: Anatomical MRI (T1-weighted) images will be analyzed using voxel-based lesion-symptom mapping (VLSM, MATLAB toolbox). Voxels will be classified as "lesioned" or "non-lesioned" in gray and white matter.
  * Behavioral measures: Performance on fast-mapping tasks (recognition scores).
  Those measurements will be aggregated : VLSM will be used to generate statistical maps of significant differences in fast-mapping recognition scores between lesioned vs. non-lesioned voxels across the T1 MRI. This method allows the evaluation of statistical relationships between specific brain lesions and behavioral deficits without requiring patient grouping by lesion site or behavioral threshold. VLSM integrates permutation testing for robust statistical inference and can analyze both discrete and graded lesions. As voxels may be located in either cortical or white matter regions, the approach enables the investigation of disconnection syndromes in addition to cortical syndromes.

SECONDARY OUTCOMES:
Performance of semantic learning | Baseline
  The performance of semantic learning during social interactions will be compared to another condition without social interactions. A correlation between the time elapsed since the brain injury and the performance on semantic learning tasks will be assessed. The effect of the localisation of the lesions (hippocampal or extra-hippocampal) will be determined.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital of Caen, Caen
  - University Hospital of Toulouse, Toulouse